CLINICAL TRIAL: NCT02377973
Title: The SKOT II Cohort - a Prospective Cohort Study of Diet and Well-being in Young Danish Children Born by Obese Mothers
Brief Title: Diet and Well-being of Young Danish Children Born by Obese Mothers
Acronym: SKOT II
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Technical University of Denmark (Other); Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor MD, University of Copenhagen
Other Study IDs: D209; H-3-2010-122 (Other: The Committees on Biomedical Research Ethics for the Capital Region of Denmark)
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Growth; Overweight; Metabolic Syndrome; Obesity
Keywords: growth,; infancy,; children,; diet,; breastfeeding; complementary feeding; early life programming; tracking; physical activity
MeSH Terms: conditions — Overweight; Metabolic Syndrome; Obesity; Breast Feeding; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, faeces, white cells, plama/serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Growth and Development: Growth and Development og healthy young children born by Obese mothers

SUMMARY:
The overall aim is to provide a detailed description of growth, development and risk factors for later disease, especially obesity and metabolic disease in infants born by obese mothers and to compare them with a group of infants born by mothers without any restriction in prepregnancy BMI (SKOT I).

DETAILED DESCRIPTION:
The SKOT II is a prospective cohort study that includes children of obese mothers with a body mass index over 30 kg/m2. These mothers were invited to SKOT II while participating in a randomised study at Hvidovre Hospital, Copenhagen. The families were invited to three examinations, when the children were 9, 18 and 36 months of age. A total of 184 children were included in 2010. The examinations and the collecting of data are designed in the same way as SKOT I, a study of healthy children born by non-obese mother. The examinations takes place at Department of Nutrition, Exercise and Sports, Frederiksberg, Denmark. Following data were collected during the examinations: Anthropometry (weight, height, age- and sex specific Z scores for body composition, triceps- and subscapularis skinfolds), background interview (e.g. infant feeding, household income, the parent's educational level, allergy and chronic diseases), blood pressure (systolic, diastolic and mean arterial pressure), faeces- and urine samples, blood samples (at 9 and 36 months of age), bio impedance (at 36 months of age), 4 day diet registration, general questionnaire (e.g. sleep, daycare, attendance and use of screen devices), psychomotor questionnaire (motoric development) and 7 day physical activity monitoring (at 36 months of age).

ELIGIBILITY:
Inclusion Criteria:

* Healthy singletons born at term (week 37-43) with no disease that could influence food intake or growth. Born by obese mother (BMI ≥ 30 kg/m2) Mothers participated in a intervention study at Hvidovre Hospital

Exclusion Criteria:

* Born preterm (before week 37) Non-Danish speaking parents. Chronic disease that is expected to influence growth or food intake.

Ages: 9 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy young Danish infants born by obese morthers, who during pregnancy were part of a intervention study at Hvidovre Hospital. In the intervention at Hvidovre Hospital study the mothers were asked to join SKOT II,
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2011-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in anthropometric measurements in periods of early childhood | 9, 18 and 36 months of age
  Composite outcome consisting of body weight, height, body mass index (BMI) and BMI z-scores, waist-, upper arm- and head circumference, skinfold thickness measured at subscapularis and triceps. Compare the changes with those observed in SKOT-I (NCT02170428)
Body composition in early childhood | 36 months of age
  Body composition is measures by bio impedance. Fat mass, fat mass index (kg/m2), fat free mass index (kg/m2) are calculated. Compare the measurements with those observed in SKOT-I (NCT02170428)
Markers of Metabolic syndrome in early life | 9 and 36 months of age
  Markers consisting of triglycerides, high lipoprotein (HDL) and glucose measured in plasma/serum, waist circumference and blood pressure. Compare the measurements with those observed in SKOT-I (NCT02170428)
Diet in periods of early life | 9, 18 and 36 months of age
  The diet is recorded using self-reported record questionnaire (7 days at 9 and 18 month, 4 days at 36 month). Compare diet with the SKOT-I cohort (NCT02170428)

SECONDARY OUTCOMES:
Breastfeeding duration in infancy and early childhood | 9, 18 and 36 months of age
  Questionnaire used for assessment of exclusive and partially breastfeeding. Compare the duration with SKOT-I cohort (NCT02170428)
Insulin like growth factor at 9 and 36 months of age | 9 and 36 months of age
  Insulin like growth factor-1 and insulin like growth factor binding protein-3 concentrations in plasma. Compare the measurements with those observed in SKOT-I (NCT02170428)
Physical activity, sedentary behavior and sleep in early childhood | 9, 18 and 36 months of age
  Physical activity and sedentary behavior measured by ActiGrafph GT3X accelerometer, recording for 24 hours in 7 days at 36 months of age. Information on outdoor activity, sedentary behavior and night sleep are collected through questionnaires at 9, 18 and 36. months of age. Compare the measurements with those observed in SKOT-I (NCT02170428)
Vitamin D status in infancy | 9 and 36 months of age
  25-hydroxyvitamin D concentrations are analysed in blood samples at 9 months of age. Compare the measurements with those observed in SKOT-I (NCT02170428)
Allergy and chronic diseases | 9 and 36 months of age
  Assessment of diseases by questionnaires. Compare frequencies with those observed in SKOT-I (NCT02170428)
Appetite hormones in infancy | 9 and 36 months of age
  Leptin and adiponectin concentrations measured from blood samples. Compare the measurements with those observed in SKOT-I (NCT02170428)
Change in gut microbiota | : 9, 18 and 36 months of age
  Microbiota in the faeces analysed using polymerase chain reaction (PCR). Compare findings with SKOT-I (NCT02170428)
Achievement of milestones | 9 and 36 months of age
  Achievement of age-specific milestones by questionnaires; WHO questionnaires at 9 and 36 months of age and Ages & Stages Questionnaires (ASQ) at 36 months of age. Compare findings with SKOT-I (NCT02170428)
Metabolomics in the urine | 9, 18 and 36 months of age
  Metabolomics analysed using urine samples. Compare findings with SKOT-I (NCT02170428)

CONTACTS AND LOCATIONS:
Overall Officials: Kim F Michaelsen, MD Professor, Principal Investigator — Faculty of Science, University of Copenhagen
Locations (1):
- Department of Human Nutrition, Faculty of Sciences, University of Copenhagen, Frederiksberg, Denmark

REFERENCES:
- See also: Study homepage — http://skot.ku.dk